CLINICAL TRIAL: NCT04348357
Title: Utilizing Telemedicine for Delivery of Postoperative Care Following Minimally-invasive Gynecologic Surgery: A Randomized Controlled Trial
Brief Title: Utilizing Telemedicine for Delivery of Postoperative Care
Acronym: Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Steven Radtke, Assistant Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E19110
Record Dates: First submitted 2020-04-07; First posted 2020-04-16 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Laparoscopic Gynecologic Surgery
MeSH Terms: interventions — Telemedicine; Office Visits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Visit (Active Comparator): Patients come to the office for a traditional postoperative visit
  Interventions: Other: Office visit
- Tele-medicine (Experimental): Patients receive postoperative care via telemedicine
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — A video-call application hosted by Texas Tech University Health Science Center El Paso and easily accessible from mobile phones or video-enabled PCs will be used (webex teams)
  Arms: Tele-medicine
Other: Office visit — Patient comes to the office to receive routine postoperative care
  Arms: Traditional Visit

SUMMARY:
The investigators propose a pilot project in which enrolled patients undergoing major gynecologic surgery will be randomized to either a traditional office postoperative visit or a telemedicine postoperative visit. The two groups will then be compared on a variety of metrics including clinical outcomes, patient satisfaction and time.

DETAILED DESCRIPTION:
Project title: Utilizing telemedicine for delivery of postoperative care following minimally-invasive gynecologic surgery: A randomized controlled trial

Principal Investigator: Steven Radtke MD FACOG Co-Investigators: Randle Umeh MD Research Associate: Martha Chavez, MPA Biostatistician: Zuber Mulla, Ph.D., Professor Affiliations: Texas Tech University Health Science Center El Paso, Paul L. Foster School of Medicine

Background:

The wide-spread use of minimally invasive techniques in gynecologic surgery has brought several tangible benefits to patients including faster-recovery times, shorter hospital stays, decreased risk of long term complications, to name a few. 1-3 Technological advances such as the development of robotic assistance have allowed to further expand the number of cases that can be performed via a minimally invasive approach.4 The shift has been such that the landscape regarding operative routes in gynecologic surgery has completely reversed, with now the majority of cases being performed laparoscopically. 5 Although much has changed intraoperatively, the surrounding structure of an operative has lagged. Specifically, preoperative and post-operative visits are still conducted in a similar way than how it was done 20 years ago. Despite leaps in technology, the field of gynecologic surgery has been slow to widely implement these advances into perioperative practice. One of the specific areas of opportunity is the postoperative visit. It is common practice in the majority of fields to have a visit with the patient approximately 2 weeks after surgery. The objective of this visit is to evaluate how the patient has been progressing, examine the wound site(s), and discuss pathology results from any specimens that were removed during the procedure.

The logistics of this visit involve blocking a time-slot in an established clinic day. The patient is required to transport herself to the clinic site. Once checked-in, there may be a waiting period before being placed in a room for the practitioner to conduct the visit. Once the visit is started, as long as there are no issues, the duration of the interaction may range on average between 3-7 minutes.

Despite these visits being short and usually straight-forward, the invested time that patients have to dedicate is substantially greater than the actual interaction with the clinician. Furthermore, because of the advantages of minimally invasive surgery, many patients have already returned to work by the time of the postoperative visit which may result in a disruption of their daily work schedule.

The ubiquitousness of high-speed internet and mobile phones have allowed for the field of telemedicine to thrive in recent years.6,7 Although wide-spread application of this modality has not been implemented in the field of gynecologic surgery, other areas such as urology and pediatrics have successfully implemented telemedicine programs, specifically for postoperative patients, yielding promising results. 8,9 The investigators propose a pilot project in which enrolled patients undergoing major gynecologic surgery will be randomized to either a traditional office postoperative visit or a telemedicine postoperative visit. The two groups will then be compared on a variety of metrics including clinical outcomes, patient satisfaction and time.

Objectives

1. Determine if there are differences in patient satisfaction between traditional postoperative visits and telemedicine postoperative visits
2. Determine the difference in time invested from the patient's side and clinicians side in order to complete the postoperative visit interaction
3. Analyze if there is a difference between groups regarding visits to the emergency department related to the surgery, delayed postoperative complications, etc.

Hypothesis Patient satisfaction will be greater in the telemedicine group. The total time invested will be decreased. There will be no difference in visits to the emergency department or unrecognized postoperative complications

ELIGIBILITY:
Inclusion criteria

* Female patients between ages 18-60
* Have access to smart-phone with video/audio and internet capabilities
* Undergoing laparoscopic gynecologic surgery that requires a postoperative visit
* Total laparoscopic hysterectomy
* Laparoscopic removal of adnexal structures
* Laparoscopic excision of endometriosis

Exclusion criteria

* Patient unwilling to participate
* The patient is unwilling to install and utilize the telemedicine app on their smartphone.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Radtke, MD, Principal Investigator — TTUHSCEP
Locations (1):
- Texas Tech University Health Scince Center El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Traditional Visit | Tele-medicine
Started | 25 | 28
Completed | 25 | 16
Not Completed | 0 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Visit | Tele-medicine | Total
Number analyzed (Participants) | 25 | 16 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (7.6) | 43.3 (8.3) | 42.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 16 | 41
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 16 | 41
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.9 (6.1) | 30.6 (6.1) | 31.4 (6.0)
Distance from clinic [Mean (Standard Deviation); unit: miles] | 12.7 (7.3) | 12.5 (6.2) | 12.6 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: PSQ-18 General Satisfaction
Description: General satisfaction component from PSQ-18 (Patient Satisfaction Questionnaire-18). Ranges from 1 to 5, with 5 being the maximum score (favorable), and 1 being the minimum score (unfavorable).
Time Frame: 1 month after surgery (1-2 weeks after postoperative visit)
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Traditional Visit | Tele-medicine
Number analyzed (Participants) | 25 | 16
score on a scale | 4.0 [4.0 to 4.5] | 4.5 [4.5 to 5.0]

2. Primary Outcome: PSQ-18 Technical Quality
Description: Technical Quality component from PSQ-18 (Patient Satisfaction Questionnaire-18). Ranges from 1 to 5, with 5 being the maximum score (favorable), and 1 being the minimum score (unfavorable)
Time Frame: 1 month after surgery (1-2 weeks after postoperative visit)
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Traditional Visit | Tele-medicine
Number analyzed (Participants) | 25 | 16
score on a scale | 4.0 [3.8 to 4.5] | 4.5 [3.9 to 5.0]

3. Primary Outcome: PSQ-18 Interpersonal Manner
Description: Interpersonal manner component from PSQ-18 (Patient Satisfaction Questionnaire-18). Ranges from 1 to 5, with 5 being the maximum score (favorable), and 1 being the minimum score (unfavorable)
Time Frame: 1 month after surgery (1-2 weeks after postoperative visit)
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Traditional Visit | Tele-medicine
Number analyzed (Participants) | 25 | 16
score on a scale | 4.0 [4.0 to 4.5] | 4.5 [4.0 to 5.0]

4. Primary Outcome: PSQ-18 Communication
Description: Communication component from PSQ-18 (Patient Satisfaction Questionnaire-18). Ranges from 1 to 5, with 5 being the maximum score (favorable), and 1 being the minimum score (unfavorable)
Time Frame: 1 month after surgery (1-2 weeks after postoperative visit)
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Traditional Visit | Tele-medicine
Number analyzed (Participants) | 25 | 16
score on a scale | 4.5 [4.0 to 4.5] | 4.5 [4.3 to 5.0]

5. Primary Outcome: PSQ-18 Time Spent With Doctor
Description: "Time spent with doctor" component from PSQ-18 (Patient Satisfaction Questionnaire-18). Ranges from 1 to 5, with 5 being the maximum score (favorable), and 1 being the minimum score (unfavorable)
Time Frame: 1 month after surgery (1-2 weeks after postoperative visit)
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Traditional Visit | Tele-medicine
Number analyzed (Participants) | 25 | 16
score on a scale | 4.0 [4.0 to 4.5] | 4.5 [4.0 to 5.0]

6. Primary Outcome: PSQ-18 Accessibility and Convenience
Description: "Accessibility and convenience" component from PSQ-18 (Patient Satisfaction Questionnaire-18). Ranges from 1 to 5, with 5 being the maximum score (favorable), and 1 being the minimum score (unfavorable)
Time Frame: 1 month after surgery (1-2 weeks after postoperative visit)
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Traditional Visit | Tele-medicine
Number analyzed (Participants) | 25 | 16
score on a scale | 4.0 [3.5 to 4.5] | 4.0 [3.6 to 4.5]

7. Secondary Outcome: Actual Visit Time
Description: Time that the actual postoperative encounter took, originally to be measured in seconds, and then rounded to the nearest minute for reporting. This is measured at the time of visit by research staff using a stop-watch.
Time Frame: Measured at the time of postoperative visit, which occurred 2-3 weeks after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Traditional Visit | Tele-medicine
Number analyzed (Participants) | 25 | 16
minutes | 9.2 (4.0) | 9.1 (2.6)

8. Secondary Outcome: Visits to Emergency Department
Description: Number of visits to the emergency department occurring after the postoperative visit, within 30 days of the surgery
Time Frame: 30 days after surgery
Measure: Number; unit: number of ER visits
Arm/Group | Traditional Visit | Tele-medicine
Number analyzed (Participants) | 25 | 16
number of ER visits | 1 | 0

9. Secondary Outcome: Phone-calls to Office
Description: Number of phone-calls made to office for postoperative complaints occurring after postoperative visit, within 30 days of the surgery
Time Frame: 30 days after surgery
Measure: Number; unit: Number of phonecalls
Arm/Group | Traditional Visit | Tele-medicine
Number analyzed (Participants) | 25 | 16
Number of phonecalls | 6 | 5

10. Secondary Outcome: Time Dedicated by Patient to Complete Visit
Description: Patient estimate of the time it took them to complete the postoperative visit, including transportation to and from the clinic (if randomized to office visit group). Measured in minutes (increments of 5)
Time Frame: 1 month after surgery (1-2 weeks after postoperative visit)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Traditional Visit | Tele-medicine
Number analyzed (Participants) | 25 | 16
minutes | 60.8 (45.8) | 14.7 (11.9)

11. Secondary Outcome: Number of Patients Who Desired to Switch Groups
Description: Participants who responded YES when asked during the final interview (1-2 weeks after postoperative visit) if they would've switched groups if given the chance.
Time Frame: 1 month after surgery (1-2 weeks after postoperative visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Visit | Tele-medicine
Number analyzed (Participants) | 25 | 16
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Traditional Visit | Tele-medicine
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/16
Other Adverse Events (participants affected / at risk) | 0/25 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT04348357/Prot_SAP_000.pdf